CLINICAL TRIAL: NCT04928716
Title: Multiple Sclerosis and Voiding Symptoms: How to Assess?
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Clinical Professor, Head of neurourology department, APHP, Tenon Hospital, Paris, France, Pierre and Marie Curie University
Other Study IDs: GRC 01 GREEN
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms; Voiding Disorders
Keywords: multiple sclerosis; Lower Urinary Tract Symptoms; voiding disorders; neurogenic bladder; urodynamics
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: voiding phase evaluation — Assessment of voiding phase in multiple sclerosis patients

SUMMARY:
In multiple Sclerosis (MS), storage and voiding symptoms are well described. Urodynamic patterns underlying storage symptoms are clearly defined, but the assessment of voiding phase in neurological diseases is a sensitive topic. The international continence society (ICS) recommended performing pressure flow studies to assess voiding phase. Assessments of sphincter relaxation and detrusor contractility during voiding phase are tough aims to achieve. Indeed, there is no consensus for the detrusor contractility assessment on women or on patients with neurogenic bladder. Similarly, assessment of sphincter during bladder filling and during the voiding phase is not included in ICS recommendations. In the end, it is the physicians who conclude from the non-formalized urodynamic data if there is a DSD or detrusor underactivity. In MS patients undergoing urodynamics, studies reported 43% DSD and 12% impaired contractility. These data should be interpreted with caution due to the variability of the assessment methods.

This study aims to describe the voiding phase of MS patients with standardized urodynamic evaluation and parameters.

This prospective observational study was conducted in a neuro-urology department of a French university hospital.

All the MS patients consulting for a first urodynamic evaluation without urinary treatment were included. Standardized urodynamic evaluation included an uroflowmetry, urethral pressure profile, two pressure-flow studies. If no detrusor contractility was observed during the pressure flow studies, cystometries with 100ml/min filling rate and ice water test were performed. Anal sphincter activity was recorded using surface electromyography electrodes.

Demographic data (age, sex), disease course of the MS, treatments, Expanded Disability Status Scale, urinary symptoms using the Urinary Symptom Profile and the Neurogenic Bladder Symptom Score were collected.

For assessment of detrusor contractility, the following parameters are reported: the bladder voiding efficiency; the projected isovolumetric pressure (PIP) or bladder contractility index (BCI); the Watts factor. For women, the investigators presented 3 more parameters the PIP1; the Valentini-besson-Nelson parameter k and an urodynamic cut-off proposed by Gammie et al. for DUA. Presence of Detrusor-sphincter dyssynergia was reported if there were a detrusor contraction concurrent with an involuntary contraction of the periurethral striated muscle.

DETAILED DESCRIPTION:
Lower urinary tract (LUT) dysfunctions are common in multiple sclerosis (MS) with almost all the patients reporting LUT symptoms at 10 years of duration of MS.LUT dysfunctions affect one patient out of ten at the time of the first neurological symptoms and negatively impact patients' quality of life.

In MS, storage and voiding symptoms are well described. Urodynamic patterns underlying storage symptoms are clearly defined, but the assessment of voiding phase in neurological diseases is a sensitive topic. The international continence society (ICS) recommended to perform pressure flow studies to assess voiding phase. In 2018, the ICS defined altered sphincter function and detrusor function during pressure flow studies in neurogenic LUT dysfunction. Three types of sphincter dysfunctions are reported: detrusor-sphincter dyssynergia (DSD) defined as "a detrusor contraction concurrent with an involuntary contraction of the urethral and/or periurethral striated muscle. Occasionally flow may be prevented altogether." , non-relaxing urethral sphincter as "a non-relaxing, obstructing urethral sphincter resulting in reduced urine flow" and delayed relaxation of the urethral sphincter as "an impaired and hindered relaxation of the sphincter during voiding attempt resulting in delay of urine flow". Regarding detrusor dysfunction during voiding phase, two types are reported: Neurogenic detrusor underactivity (DUA) defined as "a contraction of reduced strength and/or duration, resulting in prolonged bladder emptying and/or a failure to achieve complete bladder emptying within a normal time span in the setting of a clinically relevant neurologic disorder", neurogenic acontractile detrusor "is one that cannot be demonstrated to contract during urodynamic studies in the setting of a clinically relevant neurologic lesion". In studies in MS patients undergoing urodynamic testing, this classification was not used. First because these definitions are recent, secondly because assessing sphincter relaxation and detrusor contractility during voiding phase are tough aims to achieve. Indeed, there is no consensus for the detrusor contractility assessment on women or on patients with neurogenic bladder. Similarly, assessment of sphincter during bladder filling and during the voiding phase is not included in ICS recommendations. In the end, it is the physicians who conclude from the non-formalized urodynamic data if there is a DSD or detrusor underactivity. In MS patients undergoing urodynamics, studies reported 43% DSD and 12% impaired contractility. These data should be interpreted with caution due to the variability of the assessment methods.

This study aims to describe the voiding phase of MS patients with standardized urodynamic evaluation and parameters.

This prospective observational study was conducted in a neuro-urology department of a French university hospital.

All the MS patients consulting for a first urodynamic evaluation without urinary treatment were included. Standardized urodynamic evaluation included an uroflowmetry, urethral pressure profile, two pressure-flow studies. If no detrusor contractility was observed during the pressure flow studies, cystometries with 100ml/min filling rate and ice water test were performed in order to identify contractility of the detrusor. Anal sphincter activity was recorded during the urodynamic testing using surface electromyography electrodes. Urodynamic evaluation was realized in accordance with ICS recommendation.

Demographic data (age, sex), disease course of the MS, treatments, Expanded Disability Status Scale (EDSS), urinary symptoms using the Urinary Symptom Profile (USP) and the Neurogenic Bladder Symptom Score (NBSS) were collected.

Detrusor contractility assessment.

For assessment of detrusor contractility on patients with neurological disease, the following parameters are reported: (i) the bladder voiding efficiency (BVE) defined as a percentage (BVE= (voided volume/total bladder capacity) x 100) ; (ii) the projected isovolumetric pressure (PIP) or bladder contractility index (BCI) given by the formula BCI=PdetQmax + 5Qmax with a strong contractility if BCI >150, normal contractility if BCI of 100-150 and weak contractility if BCI <100 ; (iii) the Watts factor (WF) = [(Pdet + a)(vdet + b) - ab]/2π where Pdet is the detrusor pressure, vdet is the velocity of detrusor contraction, and a (25 cmH2O) and b (0.6 cm/s) are back-calculated muscle constants representing the heat of shortening and the rate of energy liberation, respectively.

For women, the investigators presented 3 more parameters (i) the PIP1= PdetQmax + Qmax ; (ii) the Valentini-besson-Nelson (VBN) parameter k (simulating detrusor force) and (iii) an urodynamic cut-off proposed by Gammie et al. for DUA with PdetQmax <20; Qmax <15, and BVE <90%.

The conclusions of the detrusor contractility assessment were reported. This conclusion was made with a double reading of the urodynamic curves: the first assessment was made by the physician who initially received the patient; a second reading of the pressure-flow studies was made in blind by CC.

Bladder outlet obstruction was assessed with the Bladder Obstruction outlet index (BOOI). Presence of Detrusor-sphincter dyssynergia was reported if there were a detrusor contraction concurrent with an involuntary contraction of the periurethral striated muscle.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis (Mc Donalds criterias 2017)
* performing an urodynamic evaluation

Exclusion Criteria:

* patients with urinary treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis consulting for a first urodynamic evaluation without urinary treatment were included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Description of the voiding phase | 1 day
  assessment of the voiding phase in multiple sclerosis patients with description of the existing parameters in urodynamic tests

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PHD, Principal Investigator — Sorbonne Université, GRC 001, GREEN Groupe de Recherche en Neuro-Urologie, AP-HP, Hôpital Tenon, F-75020, Paris, France
Locations (1):
- Department of Neuro- Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided